CLINICAL TRIAL: NCT03888261
Title: Effectiveness of Mind-Body Approaches for Three Distinct Medical Conditions: A Pragmatic Randomized Controlled Television Broadcast Experiment
Brief Title: Mind-Body Approaches for Medical Conditions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); University of Copenhagen (Other); Musculoskeletal Statistics Unit, The Parker Institute (Unknown)
Responsible Party: Principal Investigator, Lina R. Khoury, Post-doctoral Researcher, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mind-Body
Record Dates: First submitted 2019-03-11; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis; Psoriasis; Heart Failure
MeSH Terms: conditions — Arthritis, Rheumatoid; Psoriasis; Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention: (Active Comparator): Mind-body intervention (incl. Relaxation Response Resiliency Program & the Open and Calm Program)
  Interventions: Behavioral: Mind-Body Approaches for Medical Conditions
- No Intervention (No Intervention): No intervention (Study participants will receive routine clinical practice)

INTERVENTIONS:
Behavioral: Mind-Body Approaches for Medical Conditions — The intervention programme of the present trial is delivered in a group-based format (15 participants per group) and overall applies three therapeutic components:
  1. Contemplative practices
  2. Psychoeducation
  3. Dialogue, including therapist-group dialogue as well as participant-participant dialogue.
  Arms: Active Intervention:

SUMMARY:
Chronic diseases are currently the most prevalent and most costly health conditions world-wide, and morbidity is expected to increase over coming years. Factors such that increased life-expectancy and certain life style-related factors, such as smoking, high-fat diet and alcohol-consumption, are commonly associated with the increase in most of the common chronic diseases. However, more complex psychosocial factors such as depression, stress, work-related dynamics and thinking patterns are thought be associated with poor health status and impaired health related quality of life among patients with suffering from chronic physical conditions (i.e. a biopsychosocial approach). Therefore, psychosocial intervention has been suggested as a complementary treatment strategy for patients with chronic conditions.

The aim of this randomized trial is to evaluate the effectiveness of mind-body multidisciplinary rehabilitation on health-related quality of life, and disease specific endpoints in people with rheumatoid arthritis, psoriasis, or heart failure.

ELIGIBILITY:
Inclusion Criteria:

Rheumatoid arthritis:

* RA according to the 1987 revised American College of Rheumatology criteria
* Not selected on the basis of their level of activity.
* The treatment of both the RA and any other medical condition have to be stable and constant for at least three months at the time of enrolment, and no future planned changes of therapy exist at the time of inclusion.
* Oral corticosteroids, if used previously, will be allowed at a maximum prednisone dose with an equivalent of 10mg/day.

Psoriasis:

* Diagnosed plaque psoriasis for 6 months or longer
* Psoriasis medical condition have to be stable and constant for at least three months at the time of enrolment (i.e. no future planned changes of therapy exist at the time of inclusion).
* Exclusion criteria are other immune-mediated conditions requiring current systemic immunosuppressant treatment except psoriatic arthritis.

Heart Failure with reduced ejection fraction:

* Symptomatic patients (NYHA class II or III, or NYHA class IV if CRT planned at enrolment) with systolic heart failure (left ventricular ejection fraction ≤40%) will be considered eligible for enrolment.
* The qualifying left ventricular ejection fraction (measured on stable heart failure medication).

Exclusion Criteria:

* Ability to participate
* Psychopathology: Persons with severe mental illness are excluded.
* Alcohol and/ or drug abuse
* Impaired cognitive functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
WHO-Five Well-being Index | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  All participants. The WHO-5 consists of five statements. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.

SECONDARY OUTCOMES:
SF36: Physical Component Summary (PCS) | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  All participants. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
SF36: Mental Component Summary (MCS) | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  All participants. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.
Illness Perception Questionnaire | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  All participants. Every item is rated using a 0-10 response scale, a higher score reflecting a more threatening view of the illness.
Pittsburgh sleep quality index | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  All participants. The measure consists of 19 individual items, creating 7 components that produce one global score. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
High-sensitivity C-reactive protein (hs-CRP) | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  All participants. Blood sample
Mindful Attention Awareness Scale-5 | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  All participants. To score the scale, simply compute a mean of the 15 items. Higher scores reflect higher levels of dispositional mindfulness
Self-Compassion Scale | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  All participants. As a rough guide, a score of 1-2.5 for your overall self-compassion score indicates you are low in self-compassion, 2.5-3.5 indicates you are moderate, and 3.5-5.0 means you are high.
Cohen's Perceived Stress Scale | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  All participants. ► Scores ranging from 0-13 would be considered low stress. ► Scores ranging from 14-26 would be considered moderate stress. ► Scores ranging from 27-40 would be considered high perceived stress
Hospital anxiety and depression scale (HADS) | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  All participants. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal. Higher score indicates worse depression or anxiety.

OTHER OUTCOMES:
Disease activity score 28 based on C-reactive protein (DAS28-CRP) | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  Rheumatoid Arthritis.
Tender joints | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  Rheumatoid Arthritis.28 joints palpates with a 4 kg pressure. The patient state the perception on pain on a scale from 1-10 cm. A higher score indicates higher pain.
Swollen joints | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  Rheumatoid Arthritis. Assessed by a train physician.
VAS-Pain | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  Rheumatoid Arthritis. Score range from 1-100. Higher score indicates worse pain.
VAS-Patient global assessment | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  Rheumatoid Arthritis. using visual analog scale (VAS) (participant global VAS). DAS28 was calculated using following formula: DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*Patient's Global VAS+0.96. Scores ranged 1.0-9.4, where lower scores indicated less disease activity.
Psoriasis Area and Severity Index | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  Psoriasis. ASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 to 72.Higher score indicates worse psoriasis.
Physician Global Assessment (PGA) | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  Psoriasis. Scores range from 100 (extremely high functioning) to 1 (severely impaired).
Dermatology Life Quality Index (DLQI) | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  Psoriasis. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Kansas City Cardiomyopathy Questionnaire | At baseline, 10-12 weeks (1-2 weeks post-intervention), and 26 weeks from baseline
  Heart Failure with reduced ejection fraction. In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status

IPD SHARING:
Plan to Share IPD: No